CLINICAL TRIAL: NCT02993510
Title: Randomised Multi-Center Study: Microfracturing With Chondro-Gide® for the Treatment of Isolated Cartilage Defects in the Knee Project-Nr.: 10830-003
Brief Title: A Randomized Controlled Trial Comparing Chondro-Gide® to Microfracture Alone for Treatment of Knee Cartilage Defects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10830-003
Record Dates: First submitted 2016-12-02; First posted 2016-12-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Cartilage Injury; Osteochondritis Dissecans
Keywords: microfracture; enhanced marrow stimulation; articular cartilage; Autologous Matrix-Induced Chondrogenesis; Chondro-Gide®; knee surgery; AMIC
MeSH Terms: conditions — Osteochondritis Dissecans; Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- microfracture (Active Comparator): Microfracture is an arthroscopic surgical technique involving placement of microfracture penetrations within the cartilage defect to provide stem cells and growth factors from the bone marrow to aid cartilage repair
  Interventions: Procedure: Microfracture
- Microfracture with Chondro-Gide sutured (Experimental): Microfracture covered with a collagen membrane (Chondro-Gide®) using atraumatic sutures in a one-step mini-arthrotomy procedure
  Interventions: Device: Chondro-Gide sutured
- Microfracture with Chondro-Gide glued (Experimental): Microfracture covered with a collagen membrane (Chondro-Gide®) using fibrin glue in a one-step mini-arthrotomy procedure
  Interventions: Device: Chondro-Gide glued

INTERVENTIONS:
Procedure: Microfracture — Microfracture is a well-established arthroscopic surgical technique for cartilage repair which involves several systematic steps, including debridement to a stable cartilage margin, careful removal of the calcified cartilage layer, and homogeneous placement of microfracture penetrations within the cartilage defect, with resultant complete defect fill by a well-anchored clot
  Arms: microfracture
Device: Chondro-Gide sutured — Implantation of Chondro-Gide membrane using atraumatic sutures following microfracture via mini-arthrotomy
  Arms: Microfracture with Chondro-Gide sutured
Device: Chondro-Gide glued — Implantation of Chondro-Gide membrane using Fibrin glue following microfracture via mini-arthrotomy
  Arms: Microfracture with Chondro-Gide glued

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of using Chondro-Gide® collagen membrane either sutured or glued compared to microfracture alone in the treatment of symptomatic cartilage defects of the knee.

DETAILED DESCRIPTION:
* Prospective, randomized, active treatment-controlled, open-label multicenter study (up to 40 sites in the US and EU).
* All subjects that meet preoperative screening eligibility criteria will be randomized to treatment with Chondro-Gide® either sutured or glued or Microfracture alone.
* Eligible and consenting subjects are randomized in a 1:1:1 ratio using centralized randomization list to receive one of the following treatments: Group I: Microfracture alone; Group II: Microfracture covered with a Chondro-Gide® membrane glued with fibrin glue (AMIC glued); Group III: Microfracture covered with a Chondro-Gide® membrane sutured (AMIC sutured)
* All subjects will be assessed at intervals post-procedure (6 weeks, 3 months, and 1,2 and 5 years).
* Subjects will be required to follow a strict pre-specified post-surgery rehabilitation protocol specific to the defect location.
* Measures to assess effectiveness and safety will be conducted at all follow-ups.
* Safety will be assessed by the collection of adverse events at all timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 50
* One or two cartilage defects Grade III or IV according to Outerbridge classification
* Defect size between 2 and 10 cm2 (inclusive)
* Intact normal surrounding cartilage to suture the Chondro-Gide® membrane
* Informed consent
* Patient willing to fulfill a strict postoperative physiotherapy scheme

Exclusion Criteria:

* More than 2 defects
* Defects on both knees
* X-ray signs of osteoarthritis
* Bone lesion > 0.7 cm in the defect
* Knee instability, varus or valgus deformation, status after complete meniscus resection, status after mosaicplasty, patella dysplasia
* Rheumatoid, infectious disease
* Skin lesion on the operated knee
* Treatment with cartilage building medication
* Drug and alcohol abuse
* Chronic heart disease, endocrine or metabolic disease, Haemophilia A/B
* Pregnancy or lactation
* Collagen allergy
* Participation in other Trials

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2003-12; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Histological evaluation of structural repair of evaluable biopsies harvested from the core of the index lesion during arthroscopy at 2 years | 2 years post-surgery
  The macroscopically assessed integration, surface properties and extent of filling of the defect and the microscopically assessed using the International Cartilage Repair Society (ICRS) score
MRI (magnetic resonance imaging) assessment of structural repair parameters. | 6 months and 1,2 and 5 years post-surgery
  Structural repair is assessed with magnetic resonance imaging (MRI, 1.5T) by an independent and blinded radiologist, with a focus on the extent, signal intensity and surface of the defect filling, integration to adjacent cartilage, and bone marrow lesion (BML).

SECONDARY OUTCOMES:
Change from Baseline in the patient's evaluation of overall knee condition using the Modified Cincinnati Knee Rating System. | 6 months and 1,2 and 5 years post-surgery
  The Change from Baseline will be evaluated.
Change from Baseline in the patient's evaluation of pain using the Visual Analog Scale (VAS). | 6 months and 1,2 and 5 years post-surgery
  The Change from Baseline will be evaluated.
Change from Baseline in the patient's evaluation of overall knee condition using the International Cartilage Repair Society (ICRS) "Cartilage Injury Evaluation Package". | 6 months and 1,2 and 5 years post-surgery
  The Change from Baseline will be evaluated.
Adverse Events (AE) Review | 5 years post-surgery
  The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE), will be collected for all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Anders, MD, Principal Investigator — University of Regensburg
Locations (7):
- Germany (7):
  - University of Regensburg, Bad Abbach
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Giessen, Giessen
  - Orthopedikum Hamburg, Hamburg
  - Unfallklinik Hannover, Hanover
  - University of Schleswig-Holstein, Lübeck
  - Sportklinik Ravensburg, Ravensburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anders S, Volz M, Frick H, Gellissen J. A Randomized, Controlled Trial Comparing Autologous Matrix-Induced Chondrogenesis (AMIC(R)) to Microfracture: Analysis of 1- and 2-Year Follow-Up Data of 2 Centers. Open Orthop J. 2013 May 3;7:133-43. doi: 10.2174/1874325001307010133. Print 2013. PMID 23730377
- [Result] Volz M, Schaumburger J, Frick H, Grifka J, Anders S. A randomized controlled trial demonstrating sustained benefit of Autologous Matrix-Induced Chondrogenesis over microfracture at five years. Int Orthop. 2017 Apr;41(4):797-804. doi: 10.1007/s00264-016-3391-0. Epub 2017 Jan 20. PMID 28108777
- [Derived] Volz M, Schaumburger J, Gellissen J, Grifka J, Anders S. A randomized controlled trial demonstrating sustained benefit of autologous matrix-induced chondrogenesis (AMIC(R)) over microfracture: 10-year follow-up. Eur J Orthop Surg Traumatol. 2024 Jul;34(5):2429-2437. doi: 10.1007/s00590-024-03948-0. Epub 2024 Apr 17. PMID 38630297